CLINICAL TRIAL: NCT05527639
Title: Does a Kegel Exercise Program Prior to Resistance Training Reduce the Risk of Stress Urinary Incontinence?
Brief Title: Kegel Exercises Prior to Strength Training to Improvestress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Darwin University (Other)
Responsible Party: Principal Investigator, Donelle Cross, Lecturer, Charles Darwin University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CharlesDarwinU
Record Dates: First submitted 2022-08-26; First posted 2022-09-02 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: A comparative study using data from 2 separate studies. Data used for the resistance training (RT) group from a foundational single cohort that investigated impact of RT on stress urinary incontinence (SUI) in a group of women participating in a RT program who had not previously done Kegel exercises (KE). New data for the KE+RT group was from 2 consecutive studies where the women completed a program of supervised / unsupervised KE. These 19 women took part in 12 weeks of RT to compare against the KE group. The findings of two separate studies in which the effect of RT on SUI and pelvic floor muscle strength was compared between women who completed 12 weeks of RT with or without prior KE. The RT group consisted of 14 women who did not have an experience in RT or KE and completed 12 weeks of RT. Women in the KE plus RT group (n=19) completed 12 weeks of Kegel exercise under the supervision of a qualified pelvic floor specialist; then completed the identical RT program as the RT group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group during study (Other): all participants completed a 12 week strength training program consisting of warm up exercises, dead-lifts and squats. They had all completed a program of Kegel exercise prior.
  Interventions: Behavioral: strength training program
- control group during study (Other): all participants completed a 12 week strength training program consisting of warm up exercises, dead-lifts and squats
  Interventions: Behavioral: strength training program

INTERVENTIONS:
Behavioral: strength training program — 12-weeks of strength training consisting of warm ups, dead-lifts, squats and cool down exercises

SUMMARY:
This comparative pre-post intervention study investigates the feasibility and benefits of Kegel exercises amongst incontinent women, prior to commencing resistance training, to reduce the risk of stress urinary incontinence compared to a group of women without prior Kegel exercises.

DETAILED DESCRIPTION:
The aim of the study is to determine whether a program of Kegel exercises prior to a resistance training program will result in reduction of stress urinary incontinence and whether this should be prescribed to incontinent women prior to performing resistance training. It is hypothesized that performing kegel exercises prior to resistance training would improve pelvic floor muscle strength and reduces the odds of experiencing SUI during resistance training.

ELIGIBILITY:
Inclusion Criteria:

* being female
* over eighteen years of age
* suffer from stress urinary incontinence
* did not perform Kegel exercises
* had no experience in regular resistance/strength training
* completed a physical activity readiness questionnaire (PAR-Q) form.

Exclusion Criteria:

* pregnancy, breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — must be female
Enrollment: 24 (Actual)
Dates: Start 2019-05-18 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
incontinence severity index (ISI) tool | Week 0
  questionnaire for self-reported frequency and severity of urinary incontinence. the higher the score, the higher the impact of incontinence
incontinence severity index (ISI) tool | Week 12
  questionnaire for self-reported frequency and severity of urinary incontinence. the higher the score, the higher the impact of incontinence
pelvic floor muscle strength | week 0
  physiotherapist report from digital palpation and perineometry
pelvic floor muscle strength | week 12
  physiotherapist report from digital palpation and perineometry

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Darwin University, Darwin, Northern Territory, Australia